CLINICAL TRIAL: NCT06952127
Title: Pilot Study Evaluating the Feasibility and Appropriateness of a Telerehabilitation Exercise Program in People With Post-COVID-19 Sequelae: a Single-center Randomized Trial.
Brief Title: Feasibility and Preliminary Efficacy of a Group-based Telerehabilitation Program in People With Post-COVID-19 Sequelae (TEPCO).
Acronym: TEPCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre intégré universitaire de santé et de services sociaux de la Mauricie-et-du-Centre-du-Québec (Other)
Responsible Party: Principal Investigator, Marie-Claude Lehoux, Principal Investigator, Centre intégré universitaire de santé et de services sociaux de la Mauricie-et-du-Centre-du-Québec
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-667; 889 (Registry Identifier: Base de données des projets de recherche du CIUSSS-MCQ)
Record Dates: First submitted 2025-04-24; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Long COVID-19 Syndrome; Long COVID; Long COVID Syndrome
Keywords: telerehabilitation
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telerehabilitation group (Experimental): Rehabilitation program including cardiovascular, muscular and balance training and, if necessary, respiratory physiotherapy using the Teams platform supervised by a certified kinesiologist. The rehabilitation will be conducted 3 times a week for 8 weeks in group of 5 or 6 persons.
  Interventions: Other: Rehabilitation program
- Face-to-face group (Active Comparator): Rehabilitation program including cardiovascular, muscular and balance training and, if necessary, respiratory physiotherapy at the university kinesiology clinic supervised by a certified kinesiologist. The rehabilitation will be conducted 3 times a week for 8 weeks in group of 5 or 6 persons.
  Interventions: Other: Rehabilitation program

INTERVENTIONS:
Other: Rehabilitation program — * 5-minute warm-up including easy global exercises
  * 5 resistance training exercises targeting upper and lower muscle groups
  * 30 secondes break between sets
  * Cooldown with breathing and stretching exercises

SUMMARY:
The goal of this study pilot randomized controlled study is to evaluate the feasibility of the study procedures and to compare the preliminary efficacy of a rehabilitation program given in a "remote" (telerehabilitation) or "face-to-face" model for adult patients who had confirmed SARS-CoV-2 infection and still have symptoms after eight weeks of infection. The main question it aims to answer is:

* Are the study procedures feasible?
* Will the two groups have similar results for the preliminary efficacy outcomes?

Researchers will compare group telerehabilitation to a face-to-face group to see if it's comparable.

Participants will:

* Take part in a 60-minute training session, 3 times a week in person or remotely
* Visit the clinic before starting the training program and after 8 weeks of training
* Keep a diary of their symptoms, if any

ELIGIBILITY:
Inclusion Criteria:

* adult patients (≥18 years)
* confirmed SARS-CoV-2 infection defined by positive polymerase chain reaction (PCR) testing and/or antigen test results
* referred to the pneumology clinic for a modified British Medical Research Council (mMRC) dyspnea score of 2-3 after a minimum of eight weeks of infection
* VO₂max of less than 80% of the predicted value
* receiving a medical prescription for rehabilitation following initial assessment by a pulmonologist
* being able to walk independently
* providing informed consent
* having a good internet connection (i.e., a minimum download speed of 4 Mbps and an upload speed of 4 Mbps)
* being in possession of a computer or tablet equipped with a camera enabling videoconferencing.

Exclusion Criteria:

* requiring in-hospital rehabilitation at discharge
* evidence of medical instability (i.e., moderate or severe cardiac disease, ischemic or severe hemorrhagic stroke, or neurodegenerative disease, unstable fracture)
* history of severe cognitive or mental impairment
* already enrolled in another rehabilitation program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2023-04-07 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
The feasibility of study procedures | 8 weeks
  This will be evaluated by % of participants that accept to participate in the study (recruitment rate), % of participants who drop out or withdraw from a study (attrition rate), % completed session (adherence rate); number of adverse events and % of participants satisfaction.

SECONDARY OUTCOMES:
Exercise capacity | 8 weeks
  Pedaling time on a cycle ergometer at constant load (i.e., 60% of maximum load).
Walking capacity | 8 weeks
  6-minute walk test Total distance walked in meters
Lower-limb endurance | 8 weeks
  1-minute sit-to-stand test The number of completed sit-to-stand repetitions is record.
Physical performance | 8 weeks
  Short Physical Performance Battery test Is made up of a set of three tests: standing static balance in three positions (score 0-4); lower limb strength and power through getting up and sitting on a chair(score 0-4); and walking speed at normal pace (score 0-4). And an overall score on 12.
Change in Independence in activities of daily living | 8 weeks
  The Barthel Index Ten items are scored with a number of points (the scoring is as follows: 0 = unable, 1 = needs assistance/help, 2 = independent), and then a final score is calculated by summing the points awarded to each functional skill. The higher the score, the more independent the patient is.
Change in Clinical Frailty | 8 weeks
  Clinical Frailty Scale (CFS) Frailty score ranging from 1 (very fit) to 9 (terminally ill)
Change in Quality of life | 8 weeks
  Saint George's Hospital Respiratory Questionnaire (SGHRQ). Scores ranging from 0 to 100 are calculated for each component, as well as a total score that summarizes the responses to all items. A zero score indicates no impairment of quality of life, and higher scores indicate more limitations.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre hospitalier affilié universitaire régional, Trois-Rivières, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No